CLINICAL TRIAL: NCT03203837
Title: Biomarker Analyses in Hepatocellular Carcinoma Patients Treated With Therasphere®
Brief Title: Biomarker Analyses in Hepatocellular Carcinoma (HCC) Patients Treated With TheraSphere®
Status: Terminated | Type: Observational
Why Stopped: Funding Discontinued due to low accrual rate
Sponsor: Northwestern University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Robert Lewandowski, MD, Northwestern University
Other Study IDs: STU000201854
Record Dates: First submitted 2017-06-20; First posted 2017-06-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radioembolization; Y90; TheraSphere; HCC; Biomarker; Prognostic factor; Angiogenesis; Inflammatory; Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any leftover patient plasma samples collected for this study will be retained for future research which may or may not involve genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients: HCC patients treated with radioembolization. Plasma collection will be performed at 7 timepoints in relation to treatment.
  Interventions: Other: Plasma collection

INTERVENTIONS:
Other: Plasma collection — We will be collecting plasma at 7 different timepoints in hepatocellular carcinoma patients that are treated with radioembolization.

SUMMARY:
To analyze specific angiogenic, inflammatory and immune profiles in hepatocellular carcinoma patients who undergo radioembolization.

DETAILED DESCRIPTION:
Patients who have planned lobar radioembolization (TheraSphere (TS)) and consent to this study will have peripheral blood samples collected pre-TS, post-TS, 4 hours post-TS, 24 hours post-TS, 3 days post-TS, 7 days post-TS and 30 days post-TS to analyze specific angiogenic, inflammatory and immune profiles.

ELIGIBILITY:
Inclusion Criteria:

* Must have the diagnosis of HCC (biopsy or imaging criteria)
* Must have planned lobar TheraSphere treatment
* Must be able to give consent
* Must have an ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 2
* Must have a life expectancy of ≥ 3 months
* Women must not be pregnant with an acceptable contraception in premenopausal women
* Must be > 4 weeks since prior radiation
* Must be > 2 weeks since liver surgery
* Must be ≥ 2 weeks post radiosensitizing chemotherapy or > 6 weeks since prior BCNU (carmustine) or Mitomycin-C

Exclusion Criteria:

* Patients are excluded if they do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hepatocellular carcinoma who will be receiving lobar TheraSphere radioembolization.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage change in angiogenic, inflammatory and immune biomarkers | 2 years
  The percent of change at 7 different timepoints for the following biomarkers will be calculated: Ang-2, FGFb, HB-EGF, HGF, PDGF-BB, PIGF, SDF-1, VEGF, VEGFC, IFNg, IL-1a, IL-1b, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, TNFa trimer, CRP, TGFb1, EGFR, PD-1, PD-L1, CD45RA, CD127, HLA-DR, CD62L, CD3, CD8, CD197, CCR7, CD45RO, PD-L2, FOXP3, Perforin, Granzyme, TIA-1, CD14, CD107a, CD25, CD45, CD4, CD20 and CD56+16.

SECONDARY OUTCOMES:
Treatment Response- AFP | 2 years
  Alphafetoprotein will be measured in ng/mL.
Treatment Response - Imaging | 2 years
  Lesions will be measured using mRECIST.
Treatment Response- Time-to-Progression | 2 years
  Time-to-progression will be measured in days.
Treatment Response- Overall Survival | 2 years
  Overall survival will be measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lewandowski, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poon RT, Ng IO, Lau C, Zhu LX, Yu WC, Lo CM, Fan ST, Wong J. Serum vascular endothelial growth factor predicts venous invasion in hepatocellular carcinoma: a prospective study. Ann Surg. 2001 Feb;233(2):227-35. doi: 10.1097/00000658-200102000-00012. PMID 11176129
- [Background] Ng IO, Lai EC, Fan ST, Ng MM, So MK. Prognostic significance of pathologic features of hepatocellular carcinoma. A multivariate analysis of 278 patients. Cancer. 1995 Dec 15;76(12):2443-8. doi: 10.1002/1097-0142(19951215)76:123.0.co;2-f. PMID 8625069
- [Background] Finkenzeller G, Marme D, Weich HA, Hug H. Platelet-derived growth factor-induced transcription of the vascular endothelial growth factor gene is mediated by protein kinase C. Cancer Res. 1992 Sep 1;52(17):4821-3. PMID 1511446
- [Background] Stavri GT, Hong Y, Zachary IC, Breier G, Baskerville PA, Yla-Herttuala S, Risau W, Martin JF, Erusalimsky JD. Hypoxia and platelet-derived growth factor-BB synergistically upregulate the expression of vascular endothelial growth factor in vascular smooth muscle cells. FEBS Lett. 1995 Jan 30;358(3):311-5. doi: 10.1016/0014-5793(94)01458-d. PMID 7843420
- [Background] Mann CD, Neal CP, Garcea G, Manson MM, Dennison AR, Berry DP. Prognostic molecular markers in hepatocellular carcinoma: a systematic review. Eur J Cancer. 2007 Apr;43(6):979-92. doi: 10.1016/j.ejca.2007.01.004. Epub 2007 Feb 8. PMID 17291746
- [Background] Wada H, Nagano H, Yamamoto H, Yang Y, Kondo M, Ota H, Nakamura M, Yoshioka S, Kato H, Damdinsuren B, Tang D, Marubashi S, Miyamoto A, Takeda Y, Umeshita K, Nakamori S, Sakon M, Dono K, Wakasa K, Monden M. Expression pattern of angiogenic factors and prognosis after hepatic resection in hepatocellular carcinoma: importance of angiopoietin-2 and hypoxia-induced factor-1 alpha. Liver Int. 2006 May;26(4):414-23. doi: 10.1111/j.1478-3231.2006.01243.x. PMID 16629644
- [Background] Bassullu N, Turkmen I, Dayangac M, Yagiz Korkmaz P, Yasar R, Akyildiz M, Yaprak O, Tokat Y, Yuzer Y, Bulbul Dogusoy G. The Predictive and Prognostic Significance of c-erb-B2, EGFR, PTEN, mTOR, PI3K, p27, and ERCC1 Expression in Hepatocellular Carcinoma. Hepat Mon. 2012 Oct;12(10 HCC):e7492. doi: 10.5812/hepatmon.7492. Epub 2012 Oct 11. PMID 23162604
- [Background] Ito Y, Takeda T, Sakon M, Tsujimoto M, Higashiyama S, Noda K, Miyoshi E, Monden M, Matsuura N. Expression and clinical significance of erb-B receptor family in hepatocellular carcinoma. Br J Cancer. 2001 May 18;84(10):1377-83. doi: 10.1054/bjoc.2000.1580. PMID 11355950
- [Background] Tang Z, Qin L, Wang X, Zhou G, Liao Y, Weng Y, Jiang X, Lin Z, Liu K, Ye S. Alterations of oncogenes, tumor suppressor genes and growth factors in hepatocellular carcinoma: with relation to tumor size and invasiveness. Chin Med J (Engl). 1998 Apr;111(4):313-8. PMID 10374394
- [Background] Altimari A, Fiorentino M, Gabusi E, Gruppioni E, Corti B, D'Errico A, Grigioni WF. Investigation of ErbB1 and ErbB2 expression for therapeutic targeting in primary liver tumours. Dig Liver Dis. 2003 May;35(5):332-8. doi: 10.1016/s1590-8658(03)00077-x. PMID 12846405
- [Background] Lee TY, Kim KT, Han SY. Expression of ErbB receptor proteins and TGF-alpha during diethylnitrosamine-induced hepatocarcinogenesis in the rat liver. Korean J Hepatol. 2007 Mar;13(1):70-80. PMID 17380077
- [Background] Tanabe KK, Lemoine A, Finkelstein DM, Kawasaki H, Fujii T, Chung RT, Lauwers GY, Kulu Y, Muzikansky A, Kuruppu D, Lanuti M, Goodwin JM, Azoulay D, Fuchs BC. Epidermal growth factor gene functional polymorphism and the risk of hepatocellular carcinoma in patients with cirrhosis. JAMA. 2008 Jan 2;299(1):53-60. doi: 10.1001/jama.2007.65. PMID 18167406
- [Background] Thiery JP, Sleeman JP. Complex networks orchestrate epithelial-mesenchymal transitions. Nat Rev Mol Cell Biol. 2006 Feb;7(2):131-42. doi: 10.1038/nrm1835. PMID 16493418
- [Background] Okumoto K, Hattori E, Tamura K, Kiso S, Watanabe H, Saito K, Saito T, Togashi H, Kawata S. Possible contribution of circulating transforming growth factor-beta1 to immunity and prognosis in unresectable hepatocellular carcinoma. Liver Int. 2004 Feb;24(1):21-8. doi: 10.1111/j.1478-3231.2004.00882.x. PMID 15101997
- [Background] Zulehner G, Mikula M, Schneller D, van Zijl F, Huber H, Sieghart W, Grasl-Kraupp B, Waldhor T, Peck-Radosavljevic M, Beug H, Mikulits W. Nuclear beta-catenin induces an early liver progenitor phenotype in hepatocellular carcinoma and promotes tumor recurrence. Am J Pathol. 2010 Jan;176(1):472-81. doi: 10.2353/ajpath.2010.090300. Epub 2009 Dec 11. PMID 20008139
- [Background] Takayama H, LaRochelle WJ, Sharp R, Otsuka T, Kriebel P, Anver M, Aaronson SA, Merlino G. Diverse tumorigenesis associated with aberrant development in mice overexpressing hepatocyte growth factor/scatter factor. Proc Natl Acad Sci U S A. 1997 Jan 21;94(2):701-6. doi: 10.1073/pnas.94.2.701. PMID 9012848
- [Background] Tada M, Kanai F, Tanaka Y, Tateishi K, Ohta M, Asaoka Y, Seto M, Muroyama R, Fukai K, Imazeki F, Kawabe T, Yokosuka O, Omata M. Down-regulation of hedgehog-interacting protein through genetic and epigenetic alterations in human hepatocellular carcinoma. Clin Cancer Res. 2008 Jun 15;14(12):3768-76. doi: 10.1158/1078-0432.CCR-07-1181. PMID 18559595
- [Background] Salvi A, Arici B, Portolani N, Giulini SM, De Petro G, Barlati S. In vitro c-met inhibition by antisense RNA and plasmid-based RNAi down-modulates migration and invasion of hepatocellular carcinoma cells. Int J Oncol. 2007 Aug;31(2):451-60. PMID 17611703
- [Background] Lewis CE, Pollard JW. Distinct role of macrophages in different tumor microenvironments. Cancer Res. 2006 Jan 15;66(2):605-12. doi: 10.1158/0008-5472.CAN-05-4005. PMID 16423985
- [Background] Talaat RM, Esmail AA, Elwakil R, Gurgis AA, Nasr MI. Tumor necrosis factor-alpha -308G/A polymorphism and risk of hepatocellular carcinoma in hepatitis C virus-infected patients. Chin J Cancer. 2012 Jan;31(1):29-35. doi: 10.5732/cjc.011.10258. Epub 2011 Dec 23. PMID 22200181
- [Background] Jang JW, Oh BS, Kwon JH, You CR, Chung KW, Kay CS, Jung HS. Serum interleukin-6 and C-reactive protein as a prognostic indicator in hepatocellular carcinoma. Cytokine. 2012 Dec;60(3):686-93. doi: 10.1016/j.cyto.2012.07.017. Epub 2012 Aug 18. PMID 22906998
- [Background] Castell JV, Gomez-Lechon MJ, David M, Fabra R, Trullenque R, Heinrich PC. Acute-phase response of human hepatocytes: regulation of acute-phase protein synthesis by interleukin-6. Hepatology. 1990 Nov;12(5):1179-86. doi: 10.1002/hep.1840120517. PMID 1699862
- [Background] Agata Y, Kawasaki A, Nishimura H, Ishida Y, Tsubata T, Yagita H, Honjo T. Expression of the PD-1 antigen on the surface of stimulated mouse T and B lymphocytes. Int Immunol. 1996 May;8(5):765-72. doi: 10.1093/intimm/8.5.765. PMID 8671665
- [Background] Urbani S, Amadei B, Tola D, Massari M, Schivazappa S, Missale G, Ferrari C. PD-1 expression in acute hepatitis C virus (HCV) infection is associated with HCV-specific CD8 exhaustion. J Virol. 2006 Nov;80(22):11398-403. doi: 10.1128/JVI.01177-06. Epub 2006 Sep 6. PMID 16956940
- [Background] Wenjin Z, Chuanhui P, Yunle W, Lateef SA, Shusen Z. Longitudinal fluctuations in PD1 and PD-L1 expression in association with changes in anti-viral immune response in chronic hepatitis B. BMC Gastroenterol. 2012 Aug 16;12:109. doi: 10.1186/1471-230X-12-109. PMID 22894700
- [Background] Zeng Z, Shi F, Zhou L, Zhang MN, Chen Y, Chang XJ, Lu YY, Bai WL, Qu JH, Wang CP, Wang H, Lou M, Wang FS, Lv JY, Yang YP. Upregulation of circulating PD-L1/PD-1 is associated with poor post-cryoablation prognosis in patients with HBV-related hepatocellular carcinoma. PLoS One. 2011;6(9):e23621. doi: 10.1371/journal.pone.0023621. Epub 2011 Sep 1. PMID 21912640
- [Background] Boni C, Fisicaro P, Valdatta C, Amadei B, Di Vincenzo P, Giuberti T, Laccabue D, Zerbini A, Cavalli A, Missale G, Bertoletti A, Ferrari C. Characterization of hepatitis B virus (HBV)-specific T-cell dysfunction in chronic HBV infection. J Virol. 2007 Apr;81(8):4215-25. doi: 10.1128/JVI.02844-06. Epub 2007 Feb 7. PMID 17287266
- [Background] Urbani S, Amadei B, Tola D, Pedrazzi G, Sacchelli L, Cavallo MC, Orlandini A, Missale G, Ferrari C. Restoration of HCV-specific T cell functions by PD-1/PD-L1 blockade in HCV infection: effect of viremia levels and antiviral treatment. J Hepatol. 2008 Apr;48(4):548-58. doi: 10.1016/j.jhep.2007.12.014. Epub 2008 Jan 28. PMID 18280607
- [Background] Bruix J, Gores GJ, Mazzaferro V. Hepatocellular carcinoma: clinical frontiers and perspectives. Gut. 2014 May;63(5):844-55. doi: 10.1136/gutjnl-2013-306627. Epub 2014 Feb 14. PMID 24531850
- See also: Immunotherapy and Hepatocellular Carcinoma Editorial — http://www.omicsgroup.org/journals/Immunotherapy-and-Hepatocellular-Carcinoma-2167-0889.1000e108.pdf